CLINICAL TRIAL: NCT00005053
Title: Open Label Phase II Study on Glufosfamide Administered as a 60 Minute Infusion Every 3 Weeks in Advanced Pancreatic Cancer
Brief Title: Glufosfamide With or Without Hydration in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-16994P; EORTC-16994P; ASTA-D-19575-3166
Record Dates: First submitted 2000-04-06; First posted 2004-05-03 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — beta-D-glucosylisophosphoramide mustard

INTERVENTIONS:
Drug: glufosfamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Hydration with a saline solution may protect kidney cells from the side effects of chemotherapy.

PURPOSE: Randomized phase II trial to compare the effectiveness of glufosfamide with or without hydration in treating patients who have pancreatic cancer that is metastatic or cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the activity of glufosfamide as determined by objective response in patients with metastatic or inoperable locally advanced pancreatic cancer. II. Determine the response rate in this patient population after this treatment. III. Determine the duration of objective response in these patients on this treatment. IV. Determine the toxic effects of this regimen in these patients. V. Assess the impact of hydration on the toxicity profile of this treatment in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms: Arm I: Patients receive glufosfamide IV over 1 hour on day 1. Arm II: Patients receive glufosfamide as in arm I. Patients are hydrated with excess physiological saline solution 4 hours before and for 3 hours after treatment with glufosfamide. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients with an objective complete response continue treatment for a maximum of 2 courses beyond confirmation of response. Patients are followed every 6 weeks until disease progression.

PROJECTED ACCRUAL: A total of 16-32 patients (8-16 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic or inoperable locally advanced pancreatic adenocarcinoma At least 1 target lesion accurately measurable in at least 1 dimension Longest diameter at least 20 mm with conventional techniques or at least 10 mm with spiral CT scan No symptomatic brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) Alkaline phosphatase and transaminases no greater than 2.5 times ULN (no greater than 5 times ULN for liver metastases) Renal: Creatinine no greater than 1.7 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: Normal cardiac function No history of ischemic heart disease No history of congestive heart failure within the past 6 months Normal 12 lead electrocardiogram Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other prior or concurrent malignancy, except: Cone biopsied carcinoma of the cervix Adequately treated basal or squamous cell skin cancer No unstable systemic disease No active uncontrolled infection No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent prophylactic filgrastim (G-CSF) No concurrent prophylactic growth factors Chemotherapy: No prior chemotherapy for metastatic or advanced disease Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Concurrent radiotherapy allowed provided not all target lesions are in irradiated field Surgery: At least 2 weeks since prior major surgery Other: No other concurrent anticancer agents No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 1999-12; Primary Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A. Pavlidis, MD, Study Chair — University of Ioannina
Locations (15):
- Herlev Hospital - University Hospital of Copenhagen, Herlev, Denmark
- France (4):
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
- Germany (4):
  - Universitats-Krankenhaus Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Haemato-Onkologische Praxis und Tagesklinik, Munich
  - Klinikum Nurnberg, Nuremberg
- University of Ioannina, Ioannina, Greece
- Rambam Medical Center, Haifa, Israel
- Academisch Ziekenhuis der Vrije Universiteit, Amsterdam, Netherlands
- Switzerland (3):
  - Inselspital, Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - Saint Gallen, Sankt Gallen

REFERENCES:
- [Result] Briasoulis E, Pavlidis N, Terret C, Bauer J, Fiedler W, Schoffski P, Raoul JL, Hess D, Selvais R, Lacombe D, Bachmann P, Fumoleau P. Glufosfamide administered using a 1-hour infusion given as first-line treatment for advanced pancreatic cancer. A phase II trial of the EORTC-new drug development group. Eur J Cancer. 2003 Nov;39(16):2334-40. doi: 10.1016/s0959-8049(03)00629-4. PMID 14556925